CLINICAL TRIAL: NCT03762915
Title: Effect of Non-Surgical Periodontal Therapy With and Without Minocycline HCl Microspheres, 1 mg on Bacterial Load and Systemic Markers of Inflammation
Brief Title: Scaling and Root Planing (SRP) With and Without Minocycline HCl Microspheres, 1 mg
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DENT-2018-27312
Record Dates: First submitted 2018-11-28; First posted 2018-12-04 (Actual); Results first posted 2024-03-25 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: SRP; Minocycline HCl Microspheres; Biomarkers
MeSH Terms: interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- SRP with minocycline HCl microspheres (Experimental): The intervention of minocycline HCl microspheres, 1 mg will be administered in the experimental group at baseline and the three month periodontal maintenance visit.
  Interventions: Drug: minocycline HCl microspheres
- SRP without minocycline HCl microspheres (No Intervention): The control group will not have minocycline HCl microspheres, 1 mg administered.

INTERVENTIONS:
Drug: minocycline HCl microspheres — Minocycline HCl microspheres, 1 mg are approved by the Food and Drug Administration (FDA) as an adjunct to SRP procedures for reduction of pocket depth in patients with adult periodontitis.
  Other Names: Arestin
  Arms: SRP with minocycline HCl microspheres

SUMMARY:
The primary goal of this study is to investigate the qualitative and quantitative effects of scaling and root planing (SRP) with and without minocycline HCL microspheres, 1 mg on periodontal pathogens and overall bacterial load.

A randomized controlled clinical trial of a control (SRP) group and an experimental (SRP with minocycline HCl microspheres, 1 mg) group is planned.

Specific Aim 1: Evaluate the cumulative oral periodontal bacterial burden in both control and test groups over a six month period.

Specific Aim 2: Assess gingival crevicular fluid (GCF) and serum biomarkers of inflammation.

DETAILED DESCRIPTION:
A randomized controlled clinical trial of a control (SRP) group and an experimental (SRP with minocycline HCl microspheres, 1 mg) group is planned.

The intervention of minocycline HCl microspheres, 1 mg will be administered in the experimental group at baseline and the three month periodontal maintenance visit. Saliva samples, GCF, and blood serum will be collected at four time points (baseline, 1, 3, and 6 month follow up). Saliva will be analyzed for overall pathogen burden. GCF will be analyzed for Interleukin (IL)-1, IL-6, and tumor necrosis factor alpha (TNF-α). Serum will be analyzed for C-reactive protein (hsCRP), haptoglobin (Hp), hemoglobin A1c (Hgb A1c), IL-1, IL-6, and TNF-α.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female
* At least 18 years of age
* ADA Class III-IV Chronic Periodontitis
* Scaling and Root Planing (SRP) or localized SRP
* A minimum of eight sites with pockets ≥5mm with bleeding on probing (any quadrant)

Exclusion Criteria:

* Unable to comply with study protocol
* Completed treatment of Scaling and Root Planing (SRP) and/or localized SRP within the last 6 months
* Cigarette use within the last year
* ≥2 weeks of antibiotic use in the past three months. Or antibiotic use in the last six weeks.
* Pregnant, planning to become pregnant, or unsure of pregnancy status (self- reported)
* Diagnosed cardiac conditions (cardiovascular disease (CVD) or atherosclerotic vascular disease (ASVD) including coronary heart disease, cerebrovascular disease, and peripheral artery disease, myocardial infarction, stroke, stable or unstable angina, transient ischemic attack, or coronary or other arterial revascularization
* Have any uncontrolled medical condition or immunocompromised that may impact the study (uncontrolled diabetes HbA1c > 7, HIV, etc.)
* Tetracycline allergy
* Any medication that may impact periodontal conditions (Phenytoin, calcium antagonists, cyclosporin, warfarin, or NSAIDS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Arnett, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SRP With Minocycline HCl Microspheres | SRP Without Minocycline HCl Microspheres
Started | 35 | 35
Completed | 34 | 30
Not Completed | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SRP With Minocycline HCl Microspheres | SRP Without Minocycline HCl Microspheres | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.31 (16.09) | 54.29 (14.78) | 52.8 (15.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 16 | 28
  Male | 23 | 19 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race/ethnicity data was not collected for all participants
  Participants
    number analyzed (Participants) | 34 | 26 | 60
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 4 | 3 | 7
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 9 | 4 | 13
    White | 19 | 16 | 35
    More than one race | 0 | 1 | 1
    Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Bacteria Load (log10)
Description: This is log 10 of the Bacteria load measured. The lower amount of bacteria means good conditions and the higher amount of bacteria means worse conditions.
  For data analysis fixed effects terms for log10 pathogen quantity were summarized using estimated marginal means with 95% confidence intervals (CI).
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: log 10 copies/mL
Arm/Group | SRP With Minocycline HCl Microspheres | SRP Without Minocycline HCl Microspheres
Number analyzed (Participants) | 34 | 30
log 10 copies/mL | -11.3 [-16 to -6.5] | -10.9 [-16 to -5.8]

2. Primary Outcome: Bacteria Load (log10)
Description: as for outcome 1
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: log 10 copies/mL
Arm/Group | SRP With Minocycline HCl Microspheres | SRP Without Minocycline HCl Microspheres
Number analyzed (Participants) | 34 | 30
log 10 copies/mL | -10.3 [-14.8 to -5.9] | -10.7 [-15.4 to -5.9]

3. Primary Outcome: Bacteria Load (log10)
Description: as for outcome 1
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: log 10 copies/mL
Arm/Group | SRP With Minocycline HCl Microspheres | SRP Without Minocycline HCl Microspheres
Number analyzed (Participants) | 34 | 30
log 10 copies/mL | -10.3 [-15.5 to -5.2] | -9.6 [-15.0 to -4.1]

4. Other Pre Specified Outcome: Gingival Crevicular Fluid (GCF) Markers
Description: mean
Time Frame: baseline, 1, 3, and 6 months
Population: The lab had issues with the samples and couldnt use them
Arm/Group | SRP With Minocycline HCl Microspheres | SRP Without Minocycline HCl Microspheres
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Serum Markers
Description: mean C-Reactive Protein (CRP)
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | SRP With Minocycline HCl Microspheres | SRP Without Minocycline HCl Microspheres
Number analyzed (Participants) | 34 | 30
mg/L | 2.34 (2.70) | 1.81 (1.59)

6. Other Pre Specified Outcome: Serum Markers
Description: mean CRP
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | SRP With Minocycline HCl Microspheres | SRP Without Minocycline HCl Microspheres
Number analyzed (Participants) | 34 | 30
mg/L | 1.87 (2.66) | 2.09 (2.36)

7. Other Pre Specified Outcome: Serum Markers
Description: mean CRP
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | SRP With Minocycline HCl Microspheres | SRP Without Minocycline HCl Microspheres
Number analyzed (Participants) | 34 | 30
mg/L | 1.87 (2.05) | 1.89 (2.0)

8. Other Pre Specified Outcome: Serum Markers
Description: mean CRP
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | SRP With Minocycline HCl Microspheres | SRP Without Minocycline HCl Microspheres
Number analyzed (Participants) | 34 | 30
mg/L | 1.79 (2.18) | 1.60 (2.10)

9. Other Pre Specified Outcome: Glycated Hemoglobin (HbA1c)
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | SRP With Minocycline HCl Microspheres | SRP Without Minocycline HCl Microspheres
Number analyzed (Participants) | 34 | 30
percentage | 5.53 (0.48) | 5.62 (0.98)

10. Other Pre Specified Outcome: HbA1c
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | SRP With Minocycline HCl Microspheres | SRP Without Minocycline HCl Microspheres
Number analyzed (Participants) | 34 | 30
percentage | 5.62 (0.40) | 5.64 (0.93)

11. Other Pre Specified Outcome: HbA1c
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | SRP With Minocycline HCl Microspheres | SRP Without Minocycline HCl Microspheres
Number analyzed (Participants) | 34 | 30
percentage | 5.59 (0.43) | 5.65 (0.85)

12. Other Pre Specified Outcome: HbA1c
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | SRP With Minocycline HCl Microspheres | SRP Without Minocycline HCl Microspheres
Number analyzed (Participants) | 34 | 30
percentage | 5.56 (0.40) | 5.54 (0.48)

13. Other Pre Specified Outcome: Mean Haptoglobin (Hp)
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | SRP With Minocycline HCl Microspheres | SRP Without Minocycline HCl Microspheres
Number analyzed (Participants) | 34 | 30
mg/dL | 115 (41) | 115 (48)

14. Other Pre Specified Outcome: Mean Hp
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | SRP With Minocycline HCl Microspheres | SRP Without Minocycline HCl Microspheres
Number analyzed (Participants) | 34 | 30
mg/dL | 108 (35) | 110 (39)

15. Other Pre Specified Outcome: Mean Hp
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | SRP With Minocycline HCl Microspheres | SRP Without Minocycline HCl Microspheres
Number analyzed (Participants) | 34 | 30
mg/dL | 110 (36) | 114 (38)

16. Other Pre Specified Outcome: Mean Hp
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | SRP With Minocycline HCl Microspheres | SRP Without Minocycline HCl Microspheres
Number analyzed (Participants) | 34 | 30
mg/dL | 115 (40) | 110 (38)

ADVERSE EVENTS:
Time Frame: Adverse were collected for each participant for the enrollment period of 6 months. There were no reportable adverse events.
Arm/Group | SRP With Minocycline HCl Microspheres | SRP Without Minocycline HCl Microspheres
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-09-26): https://cdn.clinicaltrials.gov/large-docs/15/NCT03762915/Prot_004.pdf
  • Informed Consent Form (2020-02-24): https://cdn.clinicaltrials.gov/large-docs/15/NCT03762915/ICF_005.pdf